CLINICAL TRIAL: NCT01240525
Title: Multicenter Randomized Phase II Study to Evaluate the Efficacy of Prophylactic Transfer of CD4 Lymphocytes After T-cell Depleted Reduced Intensity HLA-Identical Sibling Transplantation for Haematological Cancers
Brief Title: Donor Lymphocyte Infusion After Stem Cell Transplant in Treating Patients With Haematological Cancers
Acronym: ProT4
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/10/0241; UCL-10/0241 (Other: Sponsor); LRF-09041 (Other Grant/Funding Number: Leukaemia & Lymphoma Research); EU-21081 (Other); CRUK-UCL-PROT4 (Other: Cancer Research UK & UCL Cancer Trials Centre)
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Myeloma; Myelodysplastic Syndrome
Keywords: graft versus host disease; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; Waldenstrom macroglobulinemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; Non-Hodgkin's lymphoma; Hodgkin's lymphoma; Chronic (Pro-)lymphocytic leukaemia; Plasma cell myeloma; Acute myeloid leukaemia; Acute lymphoblastic leukaemia; Myelodysplastic syndrome; Chronic myelomonocytic leukaemia
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin; Hodgkin Disease; Bronchiolitis Obliterans Syndrome; Leukemia, Prolymphocytic; Multiple Myeloma; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD4 DLI (Other): Patients will receive trial product manipulated CD4 DLI post transplant as trial treatment.
  Interventions: Other: CD4 DLI
- No DLI (Other): Patients will receive no DLI post transplant as trial treatment.
  Interventions: Other: No DLI

INTERVENTIONS:
Other: CD4 DLI — Patients will receive CD4 DLI between day 70 to 115 post transplant
  Arms: CD4 DLI
Other: No DLI — Patients will not receive DLI as trial treatment
  Arms: No DLI

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and melphalan, before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) that have been treated in the laboratory after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving alemtuzumab before transplant and cyclosporine after transplant, may stop this from happening.

PURPOSE: This randomized phase II trial is studying donor lymphocyte infusion after stem cell transplant in preventing cancer relapse or cancer progression in patients with follicular lymphoma, small lymphocytic non-Hodgkin lymphoma, or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effect of prophylactic transfer of donor CD4 cells after T-cell depleted reduced-intensity HLA-identical sibling transplantation upon the risk of relapse or progression in patients with haematological cancers (e.g. NHL, HL, CLL/PLL, PCM, AML, ALL, MDS or CMML depending on the disease status).

Secondary

* To evaluate the effect of prophylactic transfer of donor CD4 cells upon the risk of graft-versus-host disease (GvHD) in these patients.
* To evaluate the effect of prophylactic transfer of donor CD4 cells upon the rates of conversion to full donor chimerism in peripheral blood in these patients.
* To determine the effect of prophylactic transfer of donor CD4 cells upon immune reconstitution in these patients.
* To evaluate the impact of prophylactic transfer of donor CD4 cells upon non-relapse mortality and overall survival of these patients.

OUTLINE: This is a multicenter study.

Patients receive fludarabine IV, melphalan IV, and alemtuzumab IV as reduced intensity conditioning for T-cell depletion followed by a reduced-intensity HLA-identical sibling stem cell transplantation on day 0. Withdrawal of cyclosporine immunosuppression therapy commence at day 40 with tapering over a period of 3-4 weeks, according to the discretion of the PI. Patients are reassessed between day 70-90 post-transplantation. Patients with stable engraftment, no significant graft-versus-host disease, and no early relapse or progression are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an allogeneic CD4 donor lymphocyte infusion (DLI) at a dose of 1 x10^6 CD4 cells/kg body weight without any other medication once between day 100-120.
* Arm II: Patients receive no further treatment.

Patients undergo blood sample collection for chimerism studies and translational research.

After completion of study treatment, patients are followed up periodically for 1 years and then annually.

Peer Reviewed and Funded or Endorsed by Bloodwise.

ELIGIBILITY:
At registration (pre-transplant)

* Haematological cancer which can be ONE OF the following:

  * Non-Hodgkin's lymphoma (NHL) in CR or PR
  * Hodgkin's lymphoma (HL) in CR or PR
  * Chronic (Pro-)lymphocytic leukaemia (CLL/PLL) in CR or PR
  * Plasma cell myeloma (PCM) in CR, VGPR or PR
  * Acute myeloid leukaemia (AML) in CR
  * Acute lymphoblastic leukaemia (ALL) in CR
  * Myelodysplastic syndrome (MDS) < 10% blasts in bone marrow
  * Chronic myelomonocytic leukaemia (CMML) < 10% blasts in bone marrow
* Have undergone disease reassessment within 8 weeks prior to registration
* HLA-identical sibling transplant to be performed using one of the following reduced intensity alemtuzumab-containing conditioning regimens:

  * Fludarabine-busulphan-alemtuzumab
  * Fludarabine-melphalan-alemtuzumab
  * BCNU-etoposide-cytarabine-melphalan (BEAM)-alemtuzumab
  * CCNU-etoposide-cytarabine-melphalan (LEAM)-alemtuzumab
* Aged ≥18 years, and <70 years
* Written informed consent

Exclusion Criteria

* Women who are pregnant or breast-feeding
* Life expectancy of <8 weeks
* Currently taking part in any other interventional clinical research study (involving any IMP, ATMP or cellular therapy)
* Organ dysfunction: Creatinine >200μmol/l, Bilirubin >50μmol/l, or AST/ALT > 3x ULN

Post-transplant

* Active acute GvHD
* Prior grade II-IV GvHD
* Relapse or progressive disease
* Primary or secondary graft failure
* Other cellular therapies
* Requirement for ongoing immunosuppression

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 1 year post-transplant | during the study and end of study

SECONDARY OUTCOMES:
Proportion of patients attaining multi-lineage full donor chimerism in peripheral blood | End of study
Incidence of infection requiring inpatient treatment | during the study and end of study
Rate of reconstitution of T-cell subsets and viral-specific immunity | End of study
Cumulative incidence of non-relapse mortality at 1 year | End of study
Overall survival and non-relapse mortality | End of study
Incidence, grade, or pattern of graft-versus-host disease | during the study and end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ronjon Chakraverty, Professor, Principal Investigator — University College Hospital London; UCL Cancer Institute
Locations (11):
- United Kingdom (11):
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - University College Hospital London (UCLH), London
  - Christie Hospital, Manchester
  - Nottingham City Hospital, Nottingham
  - Royal Hallamshire Hospital, Sheffield
  - University Hospitals Southampton, Southampton

REFERENCES:
- See also: CRUK & UCL Cancer Trial Centre - coordinating centre — http://www.ctc.ucl.ac.uk/TrialDetails.aspx?TrialID=54